CLINICAL TRIAL: NCT04137848
Title: Efficacy of Osteopathic Manipulative Treatment on Postural Control in Parkinsonian Patients With Pisa Syndrome: a Pilot Randomized Placebo-controlled Trial
Brief Title: Effects of Osteopathic Manipulative Treatment on Postural Control in Parkinson's Disease/Pisa Syndrome Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ospedale Generale Di Zona Moriggia-Pelascini (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Osteopathy2019
Record Dates: First submitted 2019-10-22; First posted 2019-10-24 (Actual); Last update posted 2020-01-18 (Actual); Status verified 2020-01

CONDITIONS: Parkinson Disease and Pisa Syndrome
MeSH Terms: conditions — Parkinson Disease | interventions — Manipulation, Osteopathic

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): Osteopathic Manipulative Treatment (OMT)+ Multidisciplinary Intensive Rehabilitation Treatment (MIRT) Osteopathic Manipulative Treatment (OMT) is manipulative therapy that was performed once a week along 30 days.
  Interventions: Procedure: Osteopathic Manipulative Treatment (OMT)+ Multidisciplinary Intensive Rehabilitation Treatment (MIRT)
- Control (Sham Comparator): Sham Osteopathic Manipulative Treatment (SOMT)+ Multidisciplinary Intensive Rehabilitation Treatment (MIRT) Osteopathic Manipulative Treatment (OMT) is manipulative therapy that was performed once a week along 30 days.
  Interventions: Procedure: Sham Osteopathic Manipulative Treatment (SOMT)+ Multidisciplinary Intensive Rehabilitation Treatment (MIRT)

INTERVENTIONS:
Procedure: Osteopathic Manipulative Treatment (OMT)+ Multidisciplinary Intensive Rehabilitation Treatment (MIRT) — OMT: 4-week manual therapeutic program with a weekly session of osteopathic examination and manipulation of somatic disfunctions in ambulatory setting. MIRT: 4-week physical therapy with 4 daily sessions (1 hour each), 5days/week, in a hospital setting. The first session comprises cardiovascular warm-up activities, relaxation, muscle stretching, exercises to improve the range of motion of different joints, exercises to improve the functionality of the abdominal muscles, and postural changes in the supine position. The second session includes exercises to improve balance and gait using stabilometric platform,treadmill plus, crossover and cycloergometer. The third and fourth pertain occupational and speech therapy.
  Arms: Experimental
Procedure: Sham Osteopathic Manipulative Treatment (SOMT)+ Multidisciplinary Intensive Rehabilitation Treatment (MIRT) — SOMT: 4-week of sham osteopathic therapeutic program with a weekly session of osteopathic examination and manipulation in ambulatory setting.
  MIRT: 4-week physical therapy with 4 daily sessions (1 hour each), 5days/week, in a hospital setting. The first session comprises cardiovascular warm-up activities, relaxation, muscle stretching, exercises to improve the range of motion of different joints, exercises to improve the functionality of the abdominal muscles, and postural changes in the supine position. The second session includes exercises to improve balance and gait using stabilometric platform,treadmill plus, crossover and cycloergometer. The third and fourth pertain occupational and speech therapy.
  Arms: Control

SUMMARY:
The aim of the study is to evaluate the efficacy of osteopathic manipulations added to an intensive, multidisciplinary rehabilitative (MIRT) program on postural control of PD-PS patients.

DETAILED DESCRIPTION:
Pisa Syndrome is frequently associated with Parkinson Disease and it is characterized by a trunk lateral flexion higher than 10 degrees that is reversible with the lying position. Its pathophysiology is multifactorial, and it is probably different depending on disease onset duration. However, a relevant association between subjective visual vertical misperception and the PS involved side was recently described. Moreover, an impairment in postural control in PD-PS patients has been recognized. Nowadays, physical therapy is the standard treatment and it is proposed to ameliorate paraspinal muscle hyperactivity and balance, as showed by previews descriptive and clinical studies. Despite being physical therapy a cornerstone in PD-PS axial symptoms treatment, the therapeutic protocol for postural control in PD-PS patients is under active study.

In recent years, preliminary studies described the effects of osteopathic manipulative treatment on motor functionality and balance in PD patients in a multidisciplinary setting, which is in line with the evidence of the need of a multidisciplinary and intensive approach to achieve better outcomes. However, the effect of OMT has never been investigated in PD-PS patients. The aim of the study is to evaluate the effects of OMT on postural control of PD-PS patients undergoing the MIRT program. Literature reported the possible benefit of OMT on the balance of healthy subjects, possibly interacting with the multisensorial integration of balance. 24 PD-PS patients are enrolled and randomized in two groups. Posturography is performed to assess Eye-closed Sway Area (ECSA) at baseline and 30 days after enrolment. The investigator who perform posturography and trunk inclination assessment is kept blinded. Trunk inclination is measured with "DIERS Formetric 4D". Other variables considered in the investigation are Eye-opened sway area (EOSA), Trunk Lateral Flexion (TLF), Kyphothic Angle (KA), Unified Parkinson Disease Rating Scale (UPDRS), Six-minute Walking Test (6MWT).

ELIGIBILITY:
Inclusion Criteria:

* Pisa Syndrome and Parkinson Disease
* PS Onset < 12 months
* TLF > 10 degrees

Exclusion Criteria:

* Scoliosis or spine deformity
* Changes of PD pharmacological therapy within 3 months
* Co-morbidity with other neurological disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2015-01 (Actual); Primary Completion 2016-09 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
Eye-closed sway area (ECSA) | 1 month
  ECSA is assessed with posturography and represents the transformation of the area described by a subject's centre of pressure in eye closed standing. It is used to assess postural stability.

SECONDARY OUTCOMES:
Trunk Lateral Flexion (TLF) | 1 month
  Area described by subject's centre of posture
Kyphothic Angle (KA) | 1 month
  Biomechanical parameter to assess subject's trunk lateral tilt.
Unified Parkinson Disease Rating Scale (UPDRS) | 1 month
  Clinical scale for Parkinson Disease (min 0 points; max 199 points) where the higher scores describes worse outcomes.
Six-minute Walking Test (6MWT) | 1 month
  Functional parameter to assess physical activity reservoir of the subjects.

CONTACTS AND LOCATIONS:
Locations (1):
- Ospedale Generale di Zona Moriggia Pelascini, Gravedona, CO, Italy